CLINICAL TRIAL: NCT00745862
Title: Illness Related Distress in Women With Clinically Localized Cutaneous Melanoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-096
Record Dates: First submitted 2008-08-22; First posted 2008-09-03 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Melanoma
Keywords: Skin
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: female patients undergoing surgical treatment of cutaneous melanoma within two years of diagnosis and treatment
  Interventions: Behavioral: questionnaire on-line or if uncomfortable with a computer interface, paper copies will be provided

INTERVENTIONS:
Behavioral: questionnaire on-line or if uncomfortable with a computer interface, paper copies will be provided — This pilot study will measure illness related distress in female patients undergoing surgical treatment of cutaneous melanoma within two years of diagnosis and treatment. Areas of particular focus will be survival anxiety, family functioning/childbearing concerns, and aesthetic impact of surgery. Patients will complete a one time only set of quality of life assessments these questionnaires will take 30-45 minutes to complete.

SUMMARY:
The purpose of this study is to examine the experiences and quality of life of women who have been treated for melanoma. By quality of life, we mean how they are feeling about different aspects of their life. In this study, we are especially interested in their feelings about survival, physical appearance and any family concerns. We will administer a series of QOL questionnaires, data sheets with many questions, to get their response to measure their feelings about these issues.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinically node-negative primary cutaneous melanoma.
* Patients participating must be female
* Patients must have completed surgical treatment for melanoma at least 10 days ago and less than 2 years at the time of study entry.

Exclusion Criteria:

* Prior history of cancer with the exception of squamous or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female melanoma patients during their regularly scheduled surgical clinic appointment at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To measure illness related distress regarding survival, family planning and functioning, and aesthetic satisfaction and QOL in post-surgical female patients diagnosed with clinically localized primary cutaneous melanoma. | conclusion of study

SECONDARY OUTCOMES:
To examine the impact of illness related distress on QOL in women treated for clinically localized primary cutaneous melanoma. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sue Brady, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Atkinson TM, Noce NS, Hay J, Rafferty BT, Brady MS. Illness-related distress in women with clinically localized cutaneous melanoma. Ann Surg Oncol. 2013 Feb;20(2):675-9. doi: 10.1245/s10434-012-2635-5. Epub 2012 Sep 11. PMID 22965568
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org